CLINICAL TRIAL: NCT04556487
Title: Investigating the Psychometric Properties of the Turkish Version of Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS)
Brief Title: Turkish Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS)
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özge ÇANKAYA, Principle investigator, Hacettepe University
Other Study IDs: GO-2020
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Developmental Delay Disorder; Genetic Disease; Metabolic Disease; Congenital Disorders; Musculoskeletal Diseases
MeSH Terms: conditions — Developmental Disabilities; Genetic Diseases, Inborn; Metabolic Diseases; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: evaluation — we will evaluate the home environment of the children asking by parents

SUMMARY:
Environment which children live and grown is very important for the all development stages. In Turkey there is no measurement for home environment evaluation so our aim is to investigate the Psychometric Properties of the Turkish version of Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS) in a sample of Turkısh children.

DETAILED DESCRIPTION:
With the advances in technology and medical fields, the rate of cerebral palsy is increasing worldwide with the increase in the survival rate of preterm, low birth weight babies and neurodevelopmentally risky babies living in neonatal intensive care units.

The International Classification of Health, Function and Disability - Child and Youth version (ICF-CY), developed by the World Health Organization, provides a common language to record problems involving functions and structures of the body, restrictions of activity and participation that occur in childhood and adolescence, and related environmental factors; and It was developed to use terminology and consists of four main components: "Body Functions", "Body Structures", "Activity and Participation", "Environmental Factors". According to ICF-CY, environmental factors that have an effect on activity and participation are changeable factors. Therefore, it is stated that environmental conditions should be changed, redesigned and the child-supportive environment should be increased in order to increase the level of activity and participation in children.

Preschool children spend most of their time at home and playing games. Toys in the game environment, playmates, parental participation and attitude play a major role in the development of the child's motor and cognitive skills and social participation (6, 7). In recent years, the importance and positive effects of the enriched environment on the motor and cognitive development of babies have been emphasized in studies. Regular neuromotor evaluations and follow-up of risky babies are guiding in establishing an early intervention program. The "Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS)" scale, developed to evaluate the characteristics of the environment in which babies live, is a valid and reliable scale that is frequently used in the literature in many different areas such as hearing loss, motor developmental delay, sensory impairment, and typical development. is a scale (8-11). Translation has been done in many different languages so far. Turkish infants at risk on a scale to evaluate the home environment in Turkey within our existing information is not yet available. It is thought that the introduction of the AHEMD-IS scale into the Turkish language will give clinicians and academicians a different perspective in the evaluation of risky babies and children.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer parents who have;
* 3-18 months child/children
* All children as typically developing children, genetic disorders, metabolic disorders, neuromotor disorders etc.

Exclusion Criteria:

* Parents who refuse to participate in the study

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Volunteer parents who have;
  * 3-18 months child/children
  * All children as typically developing children, genetic disorders, metabolic disorders, neuromotor disorders etc.
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS) | 6 months
  Psychometric properties will be investigated. AHEMD-IS have 41 items with 3 section as outside and inside environment, daily activities and toys. Questions are answered in three categories: dichotomous, 4-degree likert and explanation-based. Higher scores means good environmental enrichment.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Çankaya, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Eunson P. Aetiology and epidemiology of cerebral palsy. J Paediatr Child Health. 2012;22(9):361-6.
- [Background] 2. World Health Organization. (2007). International Classification of Functioning, Disability, and Health: Children & Youth Version: ICF-CY. World Health Organization.